CLINICAL TRIAL: NCT03783715
Title: Characterization of Treatment Responses in Lymphedema
Status: Terminated | Type: Observational
Why Stopped: Study was halted due to Covid-19 pandemic and unavailability of ketoprofen.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine, Stanford University
Other Study IDs: 49078
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Ketoprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ketoprofen: Participants will take ketoprofen for six months. They will have evaluations at baseline and month 6.
  Interventions: Drug: Ketoprofen

INTERVENTIONS:
Drug: Ketoprofen — Ketoprofen 200 mg ER, taken orally, once a day for 6 months. If medication, if obtained from a compound pharmacy, dose will be 210 mg ER, taken orally once a day for 6 months.

SUMMARY:
This study is designed to investigate the treatment response of lymphedema, of the upper or lower extremity, during clinical, pharmacologic treatment of lymphedema with oral ketoprofen. Correlation of clinical responses (changes in limb volume and skin thickness) with changes in the inflammasome will help to define the molecular substrate of treatment response.

DETAILED DESCRIPTION:
Patients presenting to the Investigator's Clinic for evaluation and treatment of (upper or lower extremity) lymphedema, will be assessed for their suitability (of low risk) for medical treatment with ketoprofen. If there are no contra-indications to taking ketoprofen, after discussion of FDA warnings, including provision of a written copy of the FDA language to the patient, and with the recommendation to discuss with the primary physician-of-record, patients will be provided with a prescription for ketoprofen 200 mg daily (one capsule taken orally, once daily) or if obtained from a compound pharmacy, ketoprofen 210 mg daily (one capsule taken orally, once daily).

Participation in this study will be offered. Two study visits, at baseline and month 6 are required. Measurements (circumferential and skin thickness) and a blood sample will be taken at each study visit.

The investigators will try to determine how ketoprofen affects the body tissue by obtaining blood samples and measurements, before starting treatment and at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of acquired lymphedema
* Stage 1, 2, or 3
* 18-75 years
* Clinical use of ketoprofen for lymphedema

Exclusion Criteria:

* Active cancer, infection, bleeding tendency, inflammatory disease and/or taking anti-inflammatory or anti-leukotriene medication will be excluded.
* Pregnant or lactating females
* Inability to take ketoprofen (contra-indicated, e.g patients with known CV, GI, renal, hepatic disease).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, may interfere with interpretation of study results, and in the judgement of the investigator, would make the participation inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Investigator's Stanford Center for Lymphatic and Venous Disorders, for evaluation and treatment of their condition, lymphedema, will be assessed for their suitability for medical treatment with ketoprofen. The use of ketoprofen in these patients is predicated upon clinical presentation and evidence-based practice, not any investigational consideration of therapy.
  If there are no contra-indications to taking ketoprofen, after discussion of FDA black box warnings, including provision of a written copy of the Medication Guide for Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), approved by FDA, will be provided to the patient, and with the recommendation to discuss with the primary physician-of-record, patients will be provided with a prescription for ketoprofen. The opportunity to participate in this observational study will be presented.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Systemic Inflammatory Mediator Granulocyte Colony Stimulating Factor (G-CSF) | baseline and month 6.
  The systemic inflammatory response of G-CSF, in patients treated with Ketoprofen will be assessed with Luminex-bead inflammasome analysis at baseline and 6 months post-treatment plasma samples. G-CSF, a glycoprotein, is an inflammatory cytokine produced by endothelium and immune cells. Ketoprofen is a unique NSAID possessing dual pathways of inflammatory inhibition, blocking cyclooxygenase (COX) and arachidonate 5-lipoxygenase (5-LO). Measurement using median fluorescence intensity (MFI) will be employed.

SECONDARY OUTCOMES:
Change in Measurement of Skin Thickness | baseline and month 6.
  Caliper-measured skin thickness (mm) of upper or lower extremities, at 3 points, will be performed and recorded. Quantitative assessment of skin thickness (mm) of the affected limb at month 6 will be compared to baseline value.
Change in Limb Volume | baseline and month 6.
  Upper or lower limbs will be marked and measured at 4 cm intervals and circumferential measurements, with tape, will be performed and recorded.
  Quantitative assessment of limb volume (ml) of the affected limb at month 6 will be compared to baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, for study endpoints, will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available 12 months after completion of the last enrollment in the trial.
Access Criteria: Data access requests will be reviewed by PI and Stanford IRB. If approved, requestors will be required to sign a data use agreement (DUA).

REFERENCES:
- [Background] Rockson SG, Tian W, Jiang X, Kuznetsova T, Haddad F, Zampell J, Mehrara B, Sampson JP, Roche L, Kim J, Nicolls MR. Pilot studies demonstrate the potential benefits of antiinflammatory therapy in human lymphedema. JCI Insight. 2018 Oct 18;3(20):e123775. doi: 10.1172/jci.insight.123775. PMID 30333315
- [Background] Tian W, Rockson SG, Jiang X, Kim J, Begaye A, Shuffle EM, Tu AB, Cribb M, Nepiyushchikh Z, Feroze AH, Zamanian RT, Dhillon GS, Voelkel NF, Peters-Golden M, Kitajewski J, Dixon JB, Nicolls MR. Leukotriene B4 antagonism ameliorates experimental lymphedema. Sci Transl Med. 2017 May 10;9(389):eaal3920. doi: 10.1126/scitranslmed.aal3920. PMID 28490670
- [Background] Nakamura K, Radhakrishnan K, Wong YM, Rockson SG. Anti-inflammatory pharmacotherapy with ketoprofen ameliorates experimental lymphatic vascular insufficiency in mice. PLoS One. 2009 Dec 21;4(12):e8380. doi: 10.1371/journal.pone.0008380. PMID 20027220
- [Background] Tabibiazar R, Cheung L, Han J, Swanson J, Beilhack A, An A, Dadras SS, Rockson N, Joshi S, Wagner R, Rockson SG. Inflammatory manifestations of experimental lymphatic insufficiency. PLoS Med. 2006 Jul;3(7):e254. doi: 10.1371/journal.pmed.0030254. PMID 16834456